CLINICAL TRIAL: NCT07391371
Title: Alternate-day Versus Daily Oral Iron Therapy in Children With Iron Deficiency Anaemia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine, Mandalay (Other)
Responsible Party: Principal Investigator, Dr Zayar Kyaw Win, Senior Consultant Paediatrician, Department of Paediatrics, University of Medicine, Mandalay
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMM-13(1/2025)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron

STUDY DESIGN:
Intervention Model Description: The study is designed as an interventional, randomized, parallel-group clinical trial. Eligible children ( total 60) with iron deficiency anaemia will be randomly assigned in a 1:1 ratio to one of two intervention groups. One group will receive oral Iron (III)-hydroxide polymaltose complex administered daily, while the other group will receive the same preparation on an alternate-day schedule. Each participant will remain in their allocated group throughout the study period, with no crossover between interventions. The parallel assignment model is chosen to allow direct comparison of the efficacy, safety, and adherence between the two dosing regimens while avoiding carryover effects, which are particularly relevant in treatments affecting serum ferritin and haemoglobin levels. The primary purpose of the study is treatment, and outcomes will be assessed through clinical evaluation and laboratory measurements over the 12 weeks follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alternate-day group (Experimental): Alternate-day group receiving oral iron III polymaltose complex 3mg/kg/day
  Interventions: Drug: Alternate-day oral Iron (III)-hydroxide polymaltose complex; Drug: Iron (III)-hydroxide polymaltose complex - daily oral dosing Iron (III)-hydroxide polymaltose complex - alternate-day oral dosing
- Daily group (Experimental): Daily group receiving oral iron III polymaltose complex 3mg/kg/day
  Interventions: Drug: Alternate-day oral Iron (III)-hydroxide polymaltose complex; Drug: Iron (III)-hydroxide polymaltose complex - daily oral dosing Iron (III)-hydroxide polymaltose complex - alternate-day oral dosing

INTERVENTIONS:
Drug: Alternate-day oral Iron (III)-hydroxide polymaltose complex — The intervention uses the same oral Iron (III)-hydroxide polymaltose complex in both study arms, differing only in dosing frequency (alternate-day versus daily administration)
Drug: Iron (III)-hydroxide polymaltose complex - daily oral dosing Iron (III)-hydroxide polymaltose complex - alternate-day oral dosing — This intervention uses oral Iron (III)-hydroxide polymaltose complex, a non-ionic ferric iron preparation, administered as a liquid formulation with dosing based on body weight. This study evaluates the same iron preparation in both study arms, with the dosing frequency (daily versus alternate-day administration) as the only variable. This approach allows assessment of the impact of dosing schedule on haemoglobin response, gastrointestinal tolerability, and treatment adherence in children with iron deficiency anaemia, while minimizing confounding from formulation-related differences.

SUMMARY:
The goal of this clinical trial is to find out whether Iron (III)-hydroxide polymaltose complex (IPC) given on an alternate-day schedule works as well as daily dosing in treating iron deficiency anaemia in children. The study will also look at the safety and tolerability of IPC.

The main questions this study aims to answer are:

Does alternate-day oral IPC improve haemoglobin levels and serum ferritin level as effectively as daily oral IPC?

Does alternate-day dosing reduce gastrointestinal side effects compared to daily dosing?

Does alternate-day dosing improve treatment adherence in children?

Researchers will compare alternate-day IPC with daily IPC to determine the most effective and well-tolerated dosing schedule for children with iron deficiency anaemia.

Participants will:

Receive oral Iron (III)-hydroxide polymaltose complex either daily or on alternate days for 12 weeks treatment period

Attend regular clinic visits for clinical assessment and blood investigations

Be monitored for adverse effects, adherence to treatment, and improvement in haemoglobin and serum ferritin levels

ELIGIBILITY:
Inclusion criteria Six months to 12 years old children with iron deficiency anaemia

Exclusion criteria

1. Critically ill child
2. Children with documented chronic illnesses (e.g., known renal failure, known liver disease)
3. Children with known cases of thalassemia
4. Children with severe anaemia requiring transfusion
5. Children who received blood transfusion within the preceding 3 months

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To study alternate-day versus daily oral iron therapy in children with iron deficiency anaemia | 1 year duration
  To compare the difference in mean haemoglobin concentration, mean serum ferritin level after 12 weeks of oral iron therapy between alternate-day and daily oral iron therapy in children with iron deficiency anaemia

SECONDARY OUTCOMES:
To compare the difference in mean haemoglobin concentration, mean serum ferritin level after 12 weeks of oral iron therapy between alternate-day and daily oral iron therapy in children with iron deficiency anaemia | one year duration

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatrics ward, 300 Beeded Teaching Hospital, Mandalay, Mandalay, Mandalay Region, Burma

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR